CLINICAL TRIAL: NCT01035086
Title: The Preventive Effects of Lupin Kernel Fibre-enriched Food on Colon Cancer and Cardiovascular Diseases in Moderate Hypercholesterolemic Subjects
Brief Title: Intervention With Lupin Kernel Fibre in Hypercholesterolemic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. G. Jahreis, University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H36-08
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Hypercholesterolemia
Keywords: dietary fibre; lupin kernel fibre; bile acids; cholesterol metabolism; blood lipids; hypercholesterolemia; fibre-enriched food; moderate hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Boregine (Experimental): Intervention: Lupinus angustifolius Boregine; 25 g lupin kernel fibre per day over 4 weeks; lupin kernel fibre was incorporated in different food
  Interventions: Dietary Supplement: fabricated food
- Reference (Active Comparator): Intervention: Reference fibre (citrus fibre: Herbacel AQ Plus; Herbafood ingredients); 25 g citrus fibre per day over 4 weeks; the citrus fibre was incorporated in different food
  Interventions: Dietary Supplement: fabricated food
- Placebo (Placebo Comparator): different food without added fibre
  Interventions: Dietary Supplement: fabricated food

INTERVENTIONS:
Dietary Supplement: fabricated food — The subjects consumed a high-fibre diet containing 25 g fibre (citrus- or lupin fibre) per day and a low-fibre diet (placebo) for four weeks each. After a one-week run-in period, each volunteer had to pass all three periods (arms) in different order with a two-week wash-out period between each.
  Other Names: diet

SUMMARY:
The objective of the conducted study was to determine the efficacy of lupin kernel fibre-enriched food (Lupinus angustifolius Boregine) on prevention of risk factors for gastrointestinal or cardiovascular diseases.

DETAILED DESCRIPTION:
Dietary fibre is suspected to effect the faecal concentration and excretion of bile acids by binding the bile acids and by increasing the faecal mass. Bile acids, especially the secondary bile acids, are potential risk factors for colorectal cancer. A high bile acid-binding ability of fibre could lead to lower blood cholesterol concentrations by interrupting the enterohepatic circulation. There is evidence that the consumption of lupin kernel fibre, containing both soluble and insoluble fibre fractions, may beneficially modify bowel health.

A total of 133 subjects were recruited for this study. Sixty moderate hypercholesterolemic volunteers (total cholesterol > 5.2 mmol/L) fulfilled the selection criteria and were randomly assigned three groups. Forty-five subjects (mean age of 47 years, 34 women and 20 men) completed the double-blind, randomized crossover trial.

The subjects consumed a high-fibre diet containing 25 g fibre (citrus- or lupin fibre) per day and a low-fibre diet (placebo) for four weeks each. After baseline, each volunteer had to pass all three periods in different order with a two-week wash-out period between each.

At the end of each intervention period, subjects consumed a standardized diet for three days. Furthermore, a quantitative stool collection took place and fasting blood samples were drawn.

ELIGIBILITY:
Inclusion Criteria:

* moderate Hypercholesterolemia (total cholesterol > 5.2 mmol/L)
* age 20-75 years

Exclusion Criteria:

* intake of lipid-lowering pharmaceuticals
* intake of nutritional supplements
* allergy against legumes
* intolerance against milk protein
* pregnancy, lactation
* chronic bowel diseases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
cholesterol metabolism (blood lipids) | after 1, 5, 10 and 15 weeks

SECONDARY OUTCOMES:
general excretion parameters, neutral sterols, bile acids, short-chain fatty acids, fibre excretion, cytotoxicity, genotoxicity | after 1, 5, 10 and 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutrional Physiology
Locations (1):
- Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutrional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Fechner A, Kiehntopf M, Jahreis G. The formation of short-chain fatty acids is positively associated with the blood lipid-lowering effect of lupin kernel fiber in moderately hypercholesterolemic adults. J Nutr. 2014 May;144(5):599-607. doi: 10.3945/jn.113.186858. Epub 2014 Feb 26. PMID 24572041